CLINICAL TRIAL: NCT05662475
Title: Effect of Non-surgical Periodontal Treatment on Visfatin, fetuin-a and Sirtuin 1 Concentrations in Gingival Crevicular Fluid of Patients With Periodontitis and Type 2 Diabetes
Brief Title: Effect of Periodontal Treatment on Visfatin, fetuin-a and Sirtuin 1 of Patients With Periodontitis and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Burcu Ozkan Cetinkaya, Professor in Periodontology, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.30.2.ODM.0.20.08/462
Record Dates: First submitted 2022-12-06; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Periodontal Diseases; Type 2 Diabetes; Periodontitis
Keywords: visfatin; fetuin-A; sirtuin 1; periodontitis; type 2 diabetes; non-surgical periodontal treatment; gingival crevicular fluid
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2; Periodontitis

STUDY DESIGN:
Intervention Model Description: Sixty-six patients were randomly divided into six equal groups; group 1: systemically and periodontally healthy individuals, group 2: systemically healthy individuals with periodontitis, group 3: controlled type 2 diabetes and periodontally healthy individuals, group 4: controlled type 2 diabetes and periodontitis, group 5: uncontrolled type 2 diabetes and periodontally healthy individuals, group 6: uncontrolled type 2 diabetes and periodontitis. The study was planned as a randomized, single-blind, parallel design. Periodontal indexes were recorded clinically and the concentrations of visfatin, fetuin-A and sirtuin 1 in gingival crevicular fluid were assessed biochemically. After baseline examinations [Silness-Löe plaque index (PI), Löe-Silness gingival index (GI), probing pocket depth (PPD), clinical attachment level (CAL), bleeding on probing (BOP)], initial periodontal treatment was completed using a full-mouth treatment protocol. Data were collected at baseline and at 3 months.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- group 1: Systemically Healthy, Periodontally Healthy (n:11) (Experimental): Plaque index, gingival index, bleeding on probing index, probing pocket depth and clinical attachment level were measured at 6 sites (buccomesial, midbuccal, buccodistal, lingual/palatal mesial, midlingual/palatal, lingual/palatal distal) of each tooth to evaluate the periodontal status of the patients. On the day of examination, panoramic radiographs were taken from all patients to determine alveolar bone loss. Gingival crevicular fluid is collected from the patients. Gingival crevicular fluid samples were collected from 5 randomly selected teeth with GI=0, PI=0 and PPD ≤3. Then, each paper strip from each tooth was individually placed in sterile 0.5 ml eppendorf tubes. Eppendorf tubes were stored at -80°C. Oral hygiene education was given to each patient. Modified Bass technique was explained as a brushing technique. Interdental brush or dental floss was recommended for interdental cleaning according to the condition of the patient's interdental areas and its use was demonstrated.
  Interventions: Diagnostic Test: GCF (gingival crevicular fluid) collection
- group 2: Systemically Healthy, Periodontitis (n:11) (Experimental): Plaque index, gingival index, bleeding on probing index, probing pocket depth and clinical attachment levels were measured from 6 sites of each tooth to evaluate the periodontal status of the patients. Panoramic radiographs were taken from all patients. Vertical/horizontal bone loss on the radiographs was evaluated to determine the stage and grade of periodontitis. Gingival crevicular fluid samples were collected from the 5 periodontal pockets with the deepest PPD before and 3 months after treatment. Eppendorf tubes were stored at -80°C. Non-surgical periodontal treatments were started under local anesthesia. Oral hygiene education was given to each patient after treatment. Modified Bass technique was explained as a brushing technique. Interdental cleaning was explained. The patient was told not to use any chemical agent for plaque removal. 3 months after the treatment gingival crevicular fluid samples are collected and clinical examination parameters were measured again.
  Interventions: Diagnostic Test: GCF (gingival crevicular fluid) collection; Procedure: Non-surgical periodontal treatment completed in 24 hours
- grup 3: Controlled Type 2 Diabetes, Periodontally Healthy (n:11) (Experimental): Plaque index, gingival index, bleeding on probing index, probing pocket depth and clinical attachment level were measured at 6 sites (buccomesial, midbuccal, buccodistal, lingual/palatal mesial, midlingual/palatal, lingual/palatal distal) of each tooth to evaluate the periodontal status of the patients. On the day of examination, panoramic radiographs were taken from all patients to determine alveolar bone loss. HbA1c values were measured. Gingival crevicular fluid is collected from the patients. Gingival crevicular fluid samples were collected from 5 randomly selected teeth with GI=0, PI=0 and PPD ≤3. Then, each paper strip from each tooth was individually placed in sterile 0.5 ml eppendorf tubes. Eppendorf tubes were stored at -80°C. Oral hygiene education was given to each patient. Modified Bass technique was explained as a brushing technique. Interdental cleaning was explained.
  Interventions: Diagnostic Test: GCF (gingival crevicular fluid) collection; Diagnostic Test: HbA1c level determination in blood serum
- group 4: Controlled Type 2 Diabetes, Periodontitis (n:11) (Experimental): Plaque index, gingival index, bleeding on probing index, probing pocket depth and clinical attachment levels were measured from 6 sites of each tooth to evaluate the periodontal status of the patients. Panoramic radiographs were taken from all patients. Vertical/horizontal bone loss on the radiographs was evaluated to determine the stage and grade of periodontitis. HbA1c levels are determined. Gingival crevicular fluid samples were collected from the 5 periodontal pockets with the deepest PPD before and 3 months after treatment. Samples were stored at -80°C. Non-surgical periodontal treatments were started under local anesthesia. Oral hygiene education was given after treatment. Modified Bass technique was explained as a brushing technique. Interdental cleaning was explained. The patient was told not to use any chemical agent for plaque removal. 3 months after the treatment gingival crevicular fluid samples are collected and clinical examination parameters were measured again.
  Interventions: Diagnostic Test: GCF (gingival crevicular fluid) collection; Procedure: Non-surgical periodontal treatment completed in 24 hours; Diagnostic Test: HbA1c level determination in blood serum
- grup 5: Uncontrolled Type 2 Diabetes, Periodontally Healthy (n:11) (Experimental): Plaque index, gingival index, bleeding on probing index, probing pocket depth and clinical attachment level were measured at 6 sites (buccomesial, midbuccal, buccodistal, lingual/palatal mesial, midlingual/palatal, lingual/palatal distal) of each tooth to evaluate the periodontal status of the patients. On the day of examination, panoramic radiographs were taken from all patients to determine alveolar bone loss. HbA1c values were measured. Gingival crevicular fluid is collected from the patients. Gingival crevicular fluid samples were collected from 5 randomly selected teeth with GI=0, PI=0 and PPD ≤3. Then, each paper strip from each tooth was individually placed in sterile 0.5 ml eppendorf tubes. Eppendorf tubes were stored at -80°C. Oral hygiene education was given to each patient. Modified Bass technique was explained as a brushing technique. Interdental cleaning was explained.
  Interventions: Diagnostic Test: GCF (gingival crevicular fluid) collection; Diagnostic Test: HbA1c level determination in blood serum
- group 6: Uncontrolled Type 2 Diabetes, Periodontitis (n:11) (Experimental): Plaque index, gingival index, bleeding on probing index, probing pocket depth and clinical attachment levels were measured from 6 sites of each tooth to evaluate the periodontal status of the patients. Panoramic radiographs were taken from all patients. Vertical/horizontal bone loss on the radiographs was evaluated to determine the stage and grade of periodontitis. HbA1c levels are determined. Gingival crevicular fluid samples were collected from the 5 periodontal pockets with the deepest PPD before and 3 months after treatment. Samples were stored at -80°C. Non-surgical periodontal treatments were started under local anesthesia. Oral hygiene education was given after treatment. Modified Bass technique was explained as a brushing technique. Interdental cleaning was explained. The patient was told not to use any chemical agent for plaque removal. 3 months after the treatment gingival crevicular fluid samples are collected and clinical examination parameters were measured again.
  Interventions: Diagnostic Test: GCF (gingival crevicular fluid) collection; Procedure: Non-surgical periodontal treatment completed in 24 hours; Diagnostic Test: HbA1c level determination in blood serum

INTERVENTIONS:
Diagnostic Test: GCF (gingival crevicular fluid) collection — Prior to GCF (gingival crevicular fluid) sampling, supragingival plaque was removed by sterile curets and, after air drying, the surfaces were isolated by cotton rolls. Gingival fluid collection strips were placed in sulcus for 30s. Care was taken not to avoid mechanical trauma and strips contaminated with blood or saliva were discarded. The absorbed GCF volume was estimated by a calibrated instrument. Then, the strips were sealed into sterile tubes before freezing at -80 °C. The readings were converted to an actual volume (μl) by reference to the standard curve.
Procedure: Non-surgical periodontal treatment completed in 24 hours — After clinical periodontal parameters were recorded and GCF samples were obtained, non-surgical periodontal treatment was started under local anesthesia. All periodontal treatments were performed by a single investigator. Local infiltrative anesthesia was applied to the buccal and palatal/lingual areas of the maxilla and mandible of the patients. After anesthesia was achieved, scaler and ultrasonic tips of various thicknesses were used together to remove supragingival and subgingival hard attachments. Root surface smoothing was performed with region-specific periodontal curettes. The roughness of the surfaces was controlled using a periodontal probe. Polishing was performed. Oral hygiene education was given to each patient after treatment. Modified Bass technique was explained as a brushing technique. Interdental cleaning is explained. The patient was told not to use any chemical agent for plaque removal.
  Arms: group 2: Systemically Healthy, Periodontitis (n:11); group 4: Controlled Type 2 Diabetes, Periodontitis (n:11); group 6: Uncontrolled Type 2 Diabetes, Periodontitis (n:11)
Diagnostic Test: HbA1c level determination in blood serum — Blood samples were taken from the patients and HbA1c concentration was measured in serum.
  Arms: group 4: Controlled Type 2 Diabetes, Periodontitis (n:11); group 6: Uncontrolled Type 2 Diabetes, Periodontitis (n:11); grup 3: Controlled Type 2 Diabetes, Periodontally Healthy (n:11); grup 5: Uncontrolled Type 2 Diabetes, Periodontally Healthy (n:11)

SUMMARY:
The aim of this study is to determine the concentrations of Visfatin, Fetuin-A and Sirtuin 1 in the gingival crevicular fluid and clinical periodontal parameters in diabetic and systemically healthy individuals and to determine whether non-surgical periodontal treatment had any effect on these biomarkers and periodontal clinical parameters at the end of a 3-month follow-up period. The hypothesis of our study is that gingival crevicular fluid Visfatin, Fetuin-A and Sirtuin 1 concentrations will change with non-surgical periodontal treatment in type 2 diabetic and systemically healthy individuals and that this change will be associated with diabetes and clinical parameters.

DETAILED DESCRIPTION:
Sixty-six patients were divided into six equal groups; group 1: systemically and periodontally healthy individuals, group 2: systemically healthy individuals with periodontitis, group 3: controlled type 2 diabetes and periodontally healthy individuals, group 4: controlled type 2 diabetes and periodontitis, group 5: uncontrolled type 2 diabetes and periodontally healthy individuals, group 6: uncontrolled type 2 diabetes and periodontitis. The study was planned as a randomized, single-blind, parallel design. Periodontal clinical parameters (Silness-Löe plaque index, Löe-Silness gingival index, probing pocket depth, clinical attachment level, bleeding on probing) were recorded clinically and concentrations of visfatin, fetuin-A and sirtuin 1 in gingival crevicular fluid were assessed biochemically. After baseline examinations, periodontal treatment was completed using a nonsurgical periodontal treatment protocol completed in 24 hours. Periodontal clinical parameters and gingival crevicular fluid were recorded at baseline and 3 months after periodontal treatment. Biochemical analysis and statistical evaluation were performed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* To be over 18 years old
* No periodontal treatment in the last 6 months
* Being systemically healthy except for type 2 diabetes
* Not taking medication for any reason except type 2 diabetes
* HbA1c <7 in controlled Type 2 diabetes group
* HbA1c ≥7 in uncontrolled Type 2 diabetes group
* Not smoking or drinking alcohol

Exclusion Criteria:

* Not volunteering to participate in the study
* Under 18 years of age
* Periodontal treatment in the last 6 months
* Having any systemic disease affecting the periodontal condition
* Having used local or systemic antibiotics in the last 3 months
* Use of anti-inflammatory, steroid drugs in the last 3 months
* Taking vitamin, mineral or antioxidant supplements in the last 3 months
* Being pregnant or lactating
* Regular use of mouthwash
* Smoking or drinking alcohol

Ages: 31 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Plaque index (PI) | Baseline to 3 months after treatment
  PI was increased in all periodontitis patients with or without type 2 diabetes. Type 2 diabetes has no effect on PI in periodontitis patients. PI was reduced after non-surgical periodontal treatment (NSPT).
Gingival index (GI) | Baseline to 3 months after treatment
  GI was increased in all periodontitis patients with or without type 2 diabetes. Type 2 diabetes has no effect on GI in periodontitis patients. GI was reduced after NSPT.
Bleeding on probing index (BPI) | Baseline to 3 months after treatment
  BPI was increased in all periodontitis patients with or without type 2 diabetes. Type 2 diabetes has no effect on BPI in periodontitis patients. BPI was reduced after NSPT.
Probable pocket depth (PPD) | Baseline to 3 months after treatment
  PPD was increased in all periodontitis patients with or without type 2 diabetes. Type 2 diabetes has no effect on PPD in periodontitis patients. PPD was reduced after NSPT.
Clinical attachment level (CAL) | Baseline to 3 months after treatment
  CAL was increased in all periodontitis patients with or without type 2 diabetes. Type 2 diabetes has no effect on CAL in periodontitis patients. CAL was reduced after NSPT.
HbA1c level in blood plasma | Baseline to 3 months after treatment
  NSPT reduced HbA1c levels of patients with type 2 diabetes.
Gingival crevicular fluid (GCF) quantity | Baseline to 3 months after treatment
  The amount of gingival crevicular fluid was not affected by periodontal status in patients with Type 2 diabetes.
Visfatin concentration in GCF | Baseline to 3 months after treatment
  Visfatin concentrations in GCF were increased in all periodontitis patients. In periodontal healthy patients with Type 2 diabetes visfatin concentrations in GCF were increased. Non-surgical periodontal treatment decreased the concentration of visfatin in GCF.
Fetuin-A concentration in GCF | Baseline to 3 months after treatment
  Fetuin-A concentrations in GCF were decreased in all periodontitis patients. In periodontal healthy patients with Type 2 diabetes fetuin-A concentrations in GCF were increased. Non-surgical periodontal treatment increased the concentration of fetuin-A in GCF.
Sirtuin 1 concentration in GCF | Baseline to 3 months after treatment
  In systemic healthy individuals, periodontitis decreased the concentration of sirtuin 1 in GCF. Type 2 diabetes increased sirtuin 1 concentration in GCF. In controlled type 2 diabetes patients with periodontitis sirtuin 1 concentrations in GCF were increased. In uncontrolled type 2 diabetes patients with periodontitis sirtuin 1 concentrations in GCF were decreased. Non-surgical periodontal treatment increased the concentration of sirtuin 1 in GCF.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu OZKAN CETINKAYA, Prof., Study Director — Ondokuzmayis University, Faculty of Dentistry, Department of Periodontology, Samsun, Turkey.; Aysun AYDEMIR INAM, Dr., Principal Investigator — Ondokuzmayis University, Faculty of Dentistry, Department of Periodontology, Samsun, Turkey.; Bahattin AVCI, Prof., Study Chair — Ondokuzmayis University, Faculty of Medicine Department of Biochemistry, Samsun, Turkey.
Locations (1):
- Ondokuz Mayıs University, Faculty of Dentistry, Department of Periodontology, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No